CLINICAL TRIAL: NCT04666727
Title: The Role of Diet and the Microbiome in Inducing Somatic Mutations in Colorectal Epithelial Cells and Its Predisposition to Carcinogenesis - A Pilot Study
Brief Title: Role of Diet on the Microbiome of the Digestive System
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1148
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool, blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to learn more about how diet affects the microbiome (bacteria and microorganisms) of the digestive system. Researchers want to learn if this, in turn, has an effect on if and how people then develop colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the differences in dietary patterns among individuals reporting to be vegetarian and omnivorous.

II. To compare the difference in stool microbiome pattern in the above mentioned two groups of individuals.

III. To compare somatic mutations in colorectal epithelial cells in the above mentioned two groups of individuals.

SECONDARY OBJECTIVE:

I. To identify and characterize an association between diet, the microbiome and its genotoxic effect on the colorectal epithelial cells and predisposition to colorectal carcinogenesis.

OUTLINE:

Participants complete dietary questionnaire over 30-60 minutes and undergo collection of stool, blood, and tissue samples for analysis via sequencing and laser dissection.

ELIGIBILITY:
Inclusion Criteria:

* GROUP I: Patients presenting for a screening colonoscopy

  * GROUP I: Age of 45 and above
  * GROUP I: Strict vegetarian diet, determined by using diet history questionnaire 3.0 National Institutes of Health (NIH)
  * GROUP I: Non smoker
  * GROUP I: Ability to understand and willingness to sign an informed consent form, complete web based dietary assessment and provide stool, colonic mucosa and blood samples
  * GROUP II: Patients presenting for a screening colonoscopy
  * GROUP II: Age of 45 and above
  * GROUP II: Omnivorous diet
  * GROUP II: Non smoker
  * GROUP II: Ability to understand and willingness to sign an informed consent form, complete web based dietary assessment and provide stool, colonic mucosa and blood sample

Exclusion Criteria:

* • Current smokers (nicotine abuse only)

  * Positive family history of colon cancer or colon cancer related syndromes
  * Recent use of antibiotics in 1 month
  * History of inflammatory bowel disease, and/or radiation enteritis or colitis
  * Pregnant and breastfeeding women
  * Women of child-bearing potential who have positive urine or serum pregnancy test
  * Heavy drinker (defined as more than 14 drinks per week)
  * Currently using anti-flatulence medications, probiotics and/or fiber supplements
  * Major dietary restrictions and/or following a special diet
  * Patient with positive fecal test/symptoms

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for a screening colonoscopy at MD Anderson West Houston
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Dietary patterns | Baseline
  Will obtain estimates of dietary patterns from colonic mucosal biopsies in each group.
Microbiome composition | Baseline
  Will obtain estimates of microbiome composition from colonic mucosal biopsies in each group. Microbiome composition will be quantified using 16S profiling will be visualized across samples using stacked bar plots and principal coordinate analysis of the weighted Unifrac distances, and microbiome diversity within each sample will be quantified using the inverse-Simpson index.
Somatic mutation burden | Baseline
  Will obtain estimates of somatic mutation burden from colonic mucosal biopsies in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Anusha Thomas, MD, Principal Investigator — MD Anderson Cancer Center, Houston, Texas
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org